CLINICAL TRIAL: NCT03127787
Title: Clinical Performance Evaluation of DxN CMV Assay
Status: Terminated | Type: Observational
Why Stopped: Business decision
Sponsor: Beckman Coulter, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CMV 2.7.3.001
Record Dates: First submitted 2017-04-17; First posted 2017-04-25 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Cytomegalovirus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: Yes

GROUPS / COHORTS (1):
- CMV infected: CMV infected observational study testing using DxN CMV Assay. Study is observational and results not used to manage patient care.
  Interventions: Diagnostic Test: CMV Assay

INTERVENTIONS:
Diagnostic Test: CMV Assay — Molecular diagnostic test to detect CMV
  Other Names: DxN CMV Assay

SUMMARY:
The DxN Cytomegalovirus (CMV) assay is an in vitro diagnostic assay intended as an aid in the management of CMV-infected individuals undergoing antiviral therapy. the purpose of the study is to establish the clinical performance of the DxN CMV Assay for plasma samples in the intended use population.

DETAILED DESCRIPTION:
same as brief summary

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Must have had a kidney transplant and be evaluated for post-transplantation care
* Must have demonstrated post-transplant CMV DNAemia
* Must be eligible for and treated with anti-CMV drugs

Exclusion Criteria:

* HIV positive
* Proven ganciclovir or valganciclovir resistance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult kidney transplant recipients undergoing CMV therapy
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
virological response to therapy | 5 months
  Resolution of CMV viremia in response to therapy as defined as 2 consecutive negative results

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - UCLA, Los Angeles, California
  - NWU, Chicago, Illinois
  - IU, Indianapolis, Indiana
  - Mayo, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No